CLINICAL TRIAL: NCT00406770
Title: Bright Light Therapy for Weight Loss
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Russian Academy of Medical Sciences (Other)
Responsible Party: Outside In
Allocation: Non-Randomized | Model: Crossover | Masking: Single | Purpose: Treatment
Other Study IDs: We-Light
Record Dates: First submitted 2006-11-30; First posted 2006-12-04 (Estimated); Last update posted 2009-10-19 (Estimated); Status verified 2009-10

CONDITIONS: Obesity
Keywords: Obesity; Light therapy; Hypocaloric diet
MeSH Terms: conditions — Obesity | interventions — Phototherapy

STUDY DESIGN:
Who Masked: Investigator
Oversight: Data Monitoring Committee: No

INTERVENTIONS:
Device: Light therapy

SUMMARY:
The study investigates whether bright artificial light adds to hypocaloric diet to lose weight in obese subjects.

DETAILED DESCRIPTION:
The study is aimed to check a preliminary evidence that bright light may help to lose weight in obese people (Thor Helge Bergan, Norvay, 2002, unpublished). Subjects: aged 20-65 y, BMI > 30, non-seasonal (SPAQ score <8, no seasonal problem), in good general health, with regular sleep from 22:00-1:00 to 6:00-9:00. Study season: November-April. Placebo-controlled, single-blind, crossover. At least 1 mo between two arms; at similar phase of menstrual cycle (if present). If could not complete at the first year, the second arm is to be done the next winter. Intervention: Lightbox (4300 lux) - during one arm, deactivated ioniser - during another arm (sequential alternation upon entering the study) for 3 weeks each morning (at least 18 days) starting between 6:00-9:00. Seating distance (from the face to the device) is 41 cm, duration - 30 min. Diet: a target amount of kcal per day is calculated based on age, weight and gender (WHO), e.g. for a woman 40 y ang 80 kg it is 1502 kcal per day. Food content - is also as recommended by WHO. Food distribution over day - usual for the particular test subject but constant over sessions. Food diary is completed daily and subjects calculate kcal themselves based on a Table of kcal. Outcomes: Weight is measured during a visit to doctor a day before and day after the 3-week session, and also at home every week. Motivation and Expectation are rated by 3-point scales in a Diary, at the beginning of each session. Mood, activity and appetite are self-estimated using a VAS-like 10-points scale every week. At the end of each arm the "Easiness of dieting" scale and Adverse event(s) are completed. In the diary, there are also columns for sleep on and off times, intervention time, duration and distance, number of kcal. A target number of subjects to complete the study is 40.

ELIGIBILITY:
Inclusion Criteria:

* age 20-65 y
* BMI > 30
* non-seasonal (SPAQ score <8, no seasonal problem)
* good general health; if there is a serious chronic disease - then compensated, with a constant dose of medication(s)
* regular sleep from 22:00-1:00 to 6:00-9:00
* a wish to participate and complete the study

Exclusion Criteria:

* any acute disease during the past month
* transmeridian travel >3 time zones over the past month
* a use of medication(s) which influence body weight - during the last 2 months

Ages: 20 Years to 65 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 41 (Actual)
Dates: Start 2006-12; Primary Completion 2007-04 (Actual); Study Completion 2007-04 (Actual)

PRIMARY OUTCOMES:
weight, kg | 4 months

CONTACTS AND LOCATIONS:
Overall Officials: Konstantin V. Danilenko, MD, Principal Investigator — Institute of Internal Medicine SB RAMS

REFERENCES:
- [Derived] Danilenko KV, Mustafina SV, Pechenkina EA. Bright light for weight loss: results of a controlled crossover trial. Obes Facts. 2013;6(1):28-38. doi: 10.1159/000348549. Epub 2013 Feb 21. PMID 23429094